CLINICAL TRIAL: NCT00272090
Title: Italian Experience Trial for the Implementation of the Use of Lantus in Basal - Bolus Regimen in Type I Diabetes Mellitus Patients.
Brief Title: Insulin Glargine in Type 1 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Trial Transparency Team, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HOE901_3507
Record Dates: First submitted 2006-01-02; First posted 2006-01-04 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-06

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Glargine

INTERVENTIONS:
Drug: Insulin glargine

SUMMARY:
The primary purpose of the protocol is to demonstrate that the new regimen (insulin glargine+regular insulin ) is no worse than the reference regimen (insulin glargine+lys-pro insulin ) in reducing the incidence of severe nocturnal hypoglycemia at the end point; the secondary purpose is to compare the two study regimens as far as the glycemic control (measured by HbA1c), the daily Mean Blood Glucose (MBG) and the mean amplitude of glycemic excursion (MAGE index), calculated on the basis of Self Monitoring Blood Glugose (SMBG) data, are concerned and to verify the safety of basal insulinization with Lantus.

ELIGIBILITY:
Inclusion criteria:

* Subjects with type 1 diabetes mellitus for more than three years
* Subjects on multiple daily injection insulin therapy, basal-bolus scheme therapy
* HbA1c <= 9 % (measured by central Lab, with DCCT aligned standard method)
* Fasting C-Peptide <= 0,1nmol/L with FBG >126 mg/dl
* Body Mass Index (BMI) < 30 kg/m2
* Willingness to accept intensive insulin therapy
* Ability and willingness to perform SMBG using plasma glucose meter
* Female subjects must be postmenopausal or under adequate contraception as judged by the investigator (it may be oral contraceptives, intra-uterine device or surgical treatment) and must have a negative serum pregnancy test

Exclusion criteria:

* Diabetes other than type 1 diabetic mellitus
* Type 1 diabetic patients with total insulin dose >= 1 IU/kg/day
* Serum creatinine > 1.5 mg/dl, or history of renal transplantation or current renal dialysis
* Congestive heart failure NYHA class II
* Acute or chronic metabolic acidosis, including diabetic ketoacidosis
* Clinical evidence of active liver disease, or serum ALT/AST 2 times the upper limit of the normal range
* Hypoglycemia unawareness
* Pregnancy or lactation
* Concomitant use of β-blockers, thiazides or systemic corticosteroids
* More than one episode of severe hypoglycemia with seizure or coma during the past year
* Likelihood of requiring treatment during the study period with any anti-diabetic drug other than the study drugs
* Failure to use adequate contraception (women of current reproductive potential only)
* Known hypersensitivity to insulin glargine, or any of the excipients
* Malignancy except basal cell carcinoma within the last five years
* Long lasting (> 2 weeks) treatment with systemic glucocorticoid therapy
* Known adrenal insufficiency (interferes with hypoglycemia counter-regulation)
* Known hemoglobinopathy or chronic anemia because it may interfere with Hb1Ac determination
* History of substance or alcohol abuse within the last two years or current addiction to substances of abuse including ethanol
* History of positive HIV test or Hepatitis B/C test
* Any usage outside of the current SPC (Summary of the Product Characteristics)
* Any clinically relevant cardiovascular, hepatic, neurologic, endocrine, or other major systemic disease other than type 1 diabetic mellitus making implementation of the protocol or interpretation of the study results difficult
* History of demonstrable micro- and macro-angiopathic complications
* Pre-planned surgery during the study
* Blood donation of more than 500 ml during the previous 3 months for males or 6 months for females
* Smoker for previous 3 months
* Receipt of an experimental drug or use of an experimental device within the 30 days prior to study entry.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 489 (Actual)
Dates: Start 2002-11; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
severe nocturnal hypoglycemias will be measured throughout the study period.

SECONDARY OUTCOMES:
HbA1c will be measured at basal and 8/16 weeks after start of treatment
8 point glucose profile will be measured during last 2 weeks before each scheduled visit
severe hypoglycemias and nocturnal hypoglycemias will be measured throughout the study period.

CONTACTS AND LOCATIONS:
Overall Officials: PAIZIS GEORGES, MD, Study Director — Sanofi